CLINICAL TRIAL: NCT01389817
Title: Near-infrared Light-emitting Diode (NIR-LED) Therapy for Leber's Hereditary Optic Neuropathy (LHON)
Acronym: LHON
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to record n95 pERG peak (primary measure), as LHON subjects are unable to focus on target.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Harry T Whelan, MD, Bleser Professor of Neurology, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO14842
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Leber's Hereditary Optic Neuropathy (LHON)
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Symptomatic LHON patients. (Experimental): Study Arm 1) symptomatic LHON patients. Male and female LHON patients with treatable bilateral optic atrophy. Treat the worse of the 2 eyes if there is a measurable difference in subjective visual functions (visual acuity, peripheral vision).
  Interventions: Device: Near-infrared light-emitting diode (NIR-LED) therapy (Med Light 630 PRO (Medical Devices Inc.))
- Asymptomatic LHON mutation carriers (No Intervention): Study Arm 2) asymptomatic LHON mutation carriers. Can be male or female; have some dysfunction, with changes occurring over months. Patients in study arm 2 will not be exposed to NIR-LED, but only undergo diagnostic studies.

INTERVENTIONS:
Device: Near-infrared light-emitting diode (NIR-LED) therapy (Med Light 630 PRO (Medical Devices Inc.)) — Subjects will be exposed to light emitted from a Med Light 630 PRO (Medical Devices Inc.) at a wavelength of 630 nm (+/-15nm) with an exposure of 4 J/cm2. This is accomplished by applying the 50 mW/cm2 LED-generated light to the closed study eye for 80 seconds. Treatments involve application of the LED-generated light for 80 seconds, twice daily.
  Other Names: Med Light 630 PRO (Medical Devices Inc.)
  Arms: Symptomatic LHON patients.

SUMMARY:
The overall objective of the proposed research is to test the hypothesis that Near-infrared Light-emitting Diode (NIR-LED) therapy will stimulate mitochondrial function, attenuate oxidative stress, and improve cell survival and vision in subjects with Leber's Hereditary Optic Neuropathy (LHON).

DETAILED DESCRIPTION:
To determine the effects of short term (3 month) near-infrared light NIR-LED therapy on anatomic and functional abnormalities of LHON as assessed by a wide variety of ophthalmologic tests, including visual acuity, optical coherence tomography, pattern electroretinography (pERG) N95 retinal ganglion cell peak, fERG-PhNR (flash ERG - Photopic Negative Response), and fundus photography.

ELIGIBILITY:
Inclusion Criteria:

* Sex - male and female. Men are affected with visual loss more frequently than women, with a male predominance of ~85%. A minimum of 25% of men and 5% of women at risk for LHON experience visual loss.
* Age - 18 years or older. The onset of visual loss typically occurs between the ages of 15 and 35 years, but otherwise classic LHON has been reported in many individuals both younger and older, with a range of age at onset from 2 to 80 years.
* Diagnosis of LHON or a carrier of the gene mutation. Patient must be evaluated by molecular confirmation, with the 11778 and other mutations of Leber's Hereditary Optic Neuropathy stratified in later data analysis.
* Able & willing to provide informed consent

Exclusion Criteria:

* Has an optic nerve disease other than LHON.
* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* Participation in an investigational trial within 30 days of NIR-LED treatment that involved treatment with any drug that has not received regulatory approval at the time of study entry. (Note: subjects cannot receive another investigational drug while participating in the study during the first 6 months.)
* Major surgery within 28 days prior to participation or major surgery planned during the next 6 months. Major surgery is defined as a surgical procedure that is more extensive than fine needle biopsy/aspiration, placement of a central venous access device, removal/biopsy of a skin lesion, or placement of a peripheral venous catheter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry T Whelan, MD, Principal Investigator — Medical College of Wisconsin
Locations (3):
- United States (3):
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - The Eye Institute, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Symptomatic LHON Patients. | Asymptomatic LHON Mutation Carriers
Started | 4 | 0
Completed | 0 | 0
Not Completed | 4 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symptomatic LHON Patients. | Asymptomatic LHON Mutation Carriers | Total
Number analyzed (Participants) | 4 | 0 | 4
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 4 |  | 4
  >=65 years | 0 |  | 0
Gender [Number; unit: participants]
  Female | 0 |  | 0
  Male | 4 |  | 4
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 4 |  | 4
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: N95 Peak Via pERG and fERG -PhNR
Description: The primary comparison will be a paired comparison of pre- and post-treatment retinal ganglion cell N95 pattern electroretinogram (pERG) peaks and fERG - Photopic Negative Response (PhNR). Pairing will be done between a subject's treatment and control eye.
Time Frame: 12 months
Population: All participants were withdrawn before any data could be obtained.
Arm/Group | Symptomatic LHON Patients. | Asymptomatic LHON Mutation Carriers
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Symptomatic LHON Patients. | Asymptomatic LHON Mutation Carriers
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 0/4 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes